CLINICAL TRIAL: NCT06614374
Title: Effects of n-3 Fatty Acids on Cognitive Function, Sleep Quality, and Bone Mineral Density in Diabetic Patients: an Ancillary Study of the Precision Nutritional Management for Diabetes (PNMD) Trial
Brief Title: Fish Oil for Cognitive Function, Sleep Quality, and Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jingjing Jiao (Other)
Responsible Party: Sponsor-Investigator, Jingjing Jiao, Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RCT_N3_SUPPLE
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Decline; Sleep; Bone Mineral Density
Keywords: Fish oil; Omega-3 fatty acids; cognitive function; sleep quality; bone density
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Placebo Comparator): Subjects will receive equivalent amounts of refined olive oil daily.
  Interventions: Dietary Supplement: Refined olive oil
- Low-dose fish oil group (Experimental): Subjects will receive four fish oil and refined olive oil mixed capsules containing 1.5 g of marine n-3 PUFAs (72% EPA and 28% DHA) per day
  Interventions: Dietary Supplement: Low-dose fish oil capsules
- High-dose fish oil group (Experimental): Subjects will receive four fish oil capsules containing 3 g of marine n-3 PUFAs (72% EPA and 28% DHA) per day
  Interventions: Dietary Supplement: High-dose fish oil capsules

INTERVENTIONS:
Dietary Supplement: Low-dose fish oil capsules — Patients in the low-dose group will receive four fish-oil and refined olive oil mixed capsules containing 1.5 g of marine n-3 PUFAs per day.
  Arms: Low-dose fish oil group
Dietary Supplement: High-dose fish oil capsules — Patients in the high-dose group will receive four fish oil capsules containing 3 g of marine n-3 PUFAs (72% EPA and 28% DHA) per day.
  Arms: High-dose fish oil group
Dietary Supplement: Refined olive oil — Participants in the control group will receive 4 g refined olive oil daily
  Arms: Control group

SUMMARY:
The Precision Nutritional Management for Diabetes trial (PNMD; NCT03708887) is a randomized clinical trial in 415 diabetic patients investigating whether taking daily dietary supplements of omega-3 fatty acids (1.5 or 3 grams) improves glucose and lipid homeostasis in Chinese diabetic patients. This ancillary study is being conducted among PNMD participants and will examine whether fish oil supplements affect A) cognitive function, B) sleep quality, and C) bone mineral density. Cognitive function, sleep quality, and bone mineral density will be evaluated at baseline and post-intervention. The Mini-Mental State Exams (MMSE) will be conducted to evaluate the cognitive function of participants. The Pittsburgh Sleep Quality Index (PSQI) will be calculated through questionnaires to evaluate sleep quality. The Dual-emission X-ray Absorptiometry (DXA) will be assessed to measure the bone density.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 2 diabetes according to WHO diagnostic criteria or those on the use of diabetic medications;
* Between 40 and 75 years old (postmenopausal women);
* Have never used n-3 PUFA supplements before or have stopped using them for more than six months.

Exclusion Criteria:

* Type 1 diabetes;
* Coronary heart disease, stroke, cancer, hepatic or kidney disease;
* Pregnancy or lactation;
* Allergy to fish;
* Have participated in other clinical trials in the last three months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Baseline and 1 year
  The Dual-emission X-ray Absorptiometry (DXA) will be assessed to measure the bone mineral density at baseline and post-intervention.
Sleep quality | Baseline and 1 year
  The Pittsburgh Sleep Quality Index (PSQI) will be calculated through questionnaires to evaluate sleep quality. The Changes in sleep quality will be quantified by the difference in PSQI scores between the baseline and the conclusion of the intervention period.
Cognitive function | Baseline and 1 year
  The Mini-Mental State Exams (MMSE) will be conducted to evaluate the cognitive function of participants at both the start and end of the study. Changes in cognitive function will be quantified by the difference in MMSE scores between the baseline and the conclusion of the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Lanxi Red Cross Hospital, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided